CLINICAL TRIAL: NCT01487005
Title: Multicenter Ozone Study in Elderly Subjects
Brief Title: Cardiovascular Effects of Exposure to Ozone
Acronym: MOSES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Health Effects Institute (Other)
Collaborators: Carelon Research (Other); University of California, San Francisco (Other); University of North Carolina, Chapel Hill (Other); University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: 10-01-4
Record Dates: First submitted 2011-12-01; First posted 2011-12-07 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Cardiovascular Injury
Keywords: ozone; air pollution; vascular function; cardiac function; inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- elderly subjects: Healthy

SUMMARY:
The Multicenter Ozone Study in Elderly Subjects will investigate whether short-term exposure of elderly volunteers to ambient levels of ozone in a controlled exposure setting causes acute cardiovascular responses as assessed by changes in blood pressure, cardiac function, and systemic biomarkers of inflammation, endothelial dysfunction, and thrombosis.

DETAILED DESCRIPTION:
This multicenter study will investigate whether short-term exposure of elderly volunteers to ambient levels of O3 in a controlled exposure setting while intermittently exercising causes acute cardiovascular responses. The study is based on the suppositions that: 1) elderly people are a susceptible group for cardiovascular effects; and 2) effects are more likely with exercise.

The study will involve approximately 90 healthy volunteers aged ≥55 and ≤70 who meet strict criteria for inclusion. They will be exposed for 3 hours to clean air, 0.07 ppm O3 (near the current NAAQS), and 0.12 ppm O3 (a level measured in several locations in the US). A suite of cardiovascular and pulmonary endpoints will be measured on the day before the exposure and up to 22 hours after the exposures. The study is being conducted at three centers using a common protocol and common SOPs. Most the endpoints will be analyzed by core laboratories to reduce the variability in the results. A Data Coordination and Analysis Center will assemble all the data generated by the three centers and conduct the statistical analyses on the combined data sets.

The study has 3 main objectives:

1. To determine the relationship of altered autonomic balance (measured as changes in heart rate and heart rate variability (HRV)), cardiac arrhythmia, and repolarization and ozone exposure.
2. To identify instances of altered systemic vascular function [measured as brachial artery flow-mediated dilation (FMD)without and with nitroglycerin (NTG) when exposed to ozone.
3. To identify pro-thrombotic vascular state (measured as increase in von Willebrand factor antigen in blood - primary endpoints) when exposed to ozone.

Additional objectives include:

1. To identify any increase in micro particle-associated tissues factor (measured as number of particles and tissue factor activity) and platelet activation) in ozone exposure.
2. To identify if markers of systemic oxidative stress and inflammation and any correlation with the cardiovascular effects and degree of airway injury (measured as CC16) and airway inflammatory effects (neutrophils and cytokines in induced sputum) in ozone exposure.
3. To determine if cardiovascular effects in ozone exposure are correlated with airway inflammatory effects, but not lung function effects.

ELIGIBILITY:
Inclusion Criteria:

* males and females of all ethnic backgrounds.
* Normal spirometry (FEV1 and FVC >75% of predicted and FEV1/FVC >0.65).
* Ability to complete the exposure exercise regimen chosen to induce a ventilation rate of 15 to 17 L/min/m2 without exceeding 80% of predicted maximal heart rate.
* Normal baseline 12-lead resting ECG, and absence of significant ST depression while performing the 15-minute required level of exercise targeted for the exposure period.
* Subjects must be able to avoid certain medication supplements listed for 1 week before the exposure.

Exclusion Criteria:

* Non-English speaking.
* Including, but not limited to as ascertained by the physicians: Subjects with chronic cardiovascular (such as ischemic heart disease) or respiratory (such as asthma or COPD) disease; diabetes, or other organ or system dysfunction; cerebrovascular disease; active psychiatric disorders that would interfere with the subject's ability to understand and participate in the study. Subjects who have tested positive for a disease that affects the immune system (such as HIV, lymphoma, leukemia) or current drug or alcohol abuse (defined as having more than 3 drinks per day or being unable to abstain from alcohol for 3 days).
* Subjects with atopy or allergic rhinitis will not be excluded as long as they do not require regular treatment with antihistamines or systemic steroids.
* Ever-smokers (smoked tobacco or marijuana during the last five years, or with history of >10 pack year for tobacco or > 1 joint year for marijuana, or living with a smoker who smokes inside the house).
* Subject having plasma cotinine level > 3ng/mL.
* BMI >35 or <18 (35 is the official cut off for class 1 obesity).
* Hypertension (defined as blood pressure >140 systolic or >90diastolic) or on anti-hypertension medications other than diuretics.
* Pregnancy or nursing (breastfeeding).
* On the following medications: prednisone, statins, beta-blockers, anticoagulants, current hormonal therapy, tamoxifen. Subjects will not be asked to discontinue needed prescription medications for the purpose of this study. If any of these medications becomes necessary during the course of the study, the subjects will be excluded. Use of other medications will be considered on an individual basis.
* Subjects taking aspirin or PDE5 inhibitors must be willing to abstain from these medications during the week preceding each exposure.
* Occupational exposures (exposed to high levels of vapors, dust, gases, or fumes on an on-going basis)

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy elderly volunteers living in or around San Francisco, CA, Research Triangle Park, NC, and Rochester, NY
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Change in endothelial function | Baseline (16 hours before exposure) and 4 hours after exposure
  Brachail artey flow-mediated dilation and nitroglycerin-mediated dilation
Change in heart rate variability | Baseline (0.5 hours before exposure) and 0.2, 2, and 21.5 after exposure
  measured with Holter monitor
Change in prothrombotic vascular state | Baseline (17 hour before exposure) and 3.5 and 22 hours after exposure
  Peripheral blood samples will be taken and stored as plasma for measurement of von Willenbrand Factor antigen
Change in cardiac repolarization | Baseline (0.5 hours before exposure) and 0.2, 2, and 21.5 after exposure
  from Holter monitor

SECONDARY OUTCOMES:
Change in markers of systemic inflammation | Baseline (17 hour before exposure) and 3.5 and 22 hours after exposure
  Peripheral blood samples will be taken and stored as plasma for measurements of inflammatory markers
Change in lung function | Baseline (0.2 hours before exposure) and 0.5, 3, and 22.5 hours after exposure
  Spirometry
Lung inflammation | 22 hours after exposure
  A sputum sample will be obtained and stored for measurement of inflammatory mediators

CONTACTS AND LOCATIONS:
Overall Officials: Anne Stoddard, PhD, Principal Investigator — Carelon Research
Locations (4):
- United States (4):
  - University of California at San Francisco, San Francisco, California
  - New England Research Institutes, Inc., Watertown, Massachusetts
  - University of Rochester, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina

REFERENCES:
- [Derived] Rich DQ, Thurston SW, Balmes JR, Bromberg PA, Arjomandi M, Hazucha MJ, Alexis NE, Ganz P, Zareba W, Thevenet-Morrison K, Koutrakis P, Frampton MW. Do Ambient Ozone or Other Pollutants Modify Effects of Controlled Ozone Exposure on Pulmonary Function? Ann Am Thorac Soc. 2020 May;17(5):563-572. doi: 10.1513/AnnalsATS.201908-597OC. PMID 32125874
- [Derived] Arjomandi M, Balmes JR, Frampton MW, Bromberg P, Rich DQ, Stark P, Alexis NE, Costantini M, Hollenbeck-Pringle D, Dagincourt N, Hazucha MJ. Respiratory Responses to Ozone Exposure. MOSES (The Multicenter Ozone Study in Older Subjects). Am J Respir Crit Care Med. 2018 May 15;197(10):1319-1327. doi: 10.1164/rccm.201708-1613OC. PMID 29232153